CLINICAL TRIAL: NCT06853899
Title: A Clinical Trial to Evaluate the Efficacy of Skin Products to Improve Skin Quality and Health
Brief Title: Clinical Trial to Evaluate the Efficacy of Skin Products to Improve Skin Quality and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truology (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20455
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Skin Hydration; Skin Aging
Keywords: Skin Quality; Facial Skin Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Truology Skincare Routine (Experimental): A single-arm study in which all participants will use the Truology Skincare Routine for 6 weeks.
  Interventions: Dietary Supplement: Truology A2; Dietary Supplement: Truology C-Boost; Dietary Supplement: Truology Barrier Restore

INTERVENTIONS:
Dietary Supplement: Truology A2 — Truology A2 (0.2% Retinaldehyde Serum) - Applied once daily at night after cleansing.
Dietary Supplement: Truology C-Boost — Truology C-Boost - Applied twice daily (morning & night).
Dietary Supplement: Truology Barrier Restore — Applied twice daily (morning & night) as the final skincare step.

SUMMARY:
This clinical trial evaluates the efficacy of three skincare products-Truology A2 (0.2% Retinaldehyde Serum), Truology C-Boost, and Truology Barrier Restore-in improving skin quality and health. The study will assess improvements in skin firmness, evenness, brightness, hydration, fine lines/wrinkles, redness, and skin stress/irritation.

ELIGIBILITY:
Inclusion Criteria:

* Be female-at-birth
* Be aged 35-55
* Anyone currently experiencing issues with skin health, including: Poor skin texture, Skin discoloration, Appearance of fine lines and wrinkles Dull skin, Poor skin firmness, Dry skin, Skin redness, Irritated and stressed skin
* Willing to use the test products as follows: Truology A2 - Once a day at night. Use 1 pump for the whole face. Use first after cleansing the skin on dry skin. C-Boost - Twice a day (AM & PM). In the morning, first use one pump for the full face after cleansing the skin. At night, use the A2 first, then C-Boost. Barrier Restore - Twice a day (AM & PM). Use one pump for the full face. Use it after C-Boost for the final step in the skincare routine, and complete questionnaires and take photos
* Have been using the same skincare routine for at least one month prior to the study, i.e., cleanser, toner, and make-up remover
* Willing to maintain the same skincare routine and products throughout the 6-week trial, e.g., moisturizer, cleanser, or SPF
* Have been consistently taking medications, oral supplements, or herbal remedies targeted at skin health and appearance for at least 3 months prior to the study and willing to maintain this routine for the duration of the study
* Agree to avoid using any other products or new forms of regular medication or supplements that target skin health and appearance
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease
* Anyone who is currently using or has used the past, exfoliating acids (AHAs/BHA) or retinoids in (i.e., salicylic acid, glycolic acid, mandelic acid, or lactic acid).
* Anyone willing to stop using exfoliating acids or retinoids for the duration of the study
* Anyone in good general health
* Anyone who resides in the United States

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Anyone currently using a prescription skin treatment
* Anyone with known severe allergic reactions
* Anyone unwilling to avoid excessive sun exposure
* Any women who are pregnant, breastfeeding, or attempting to conceive
* Anyone unwilling to follow the study protocol
* Anyone who identifies as having sensitive skin
* Anyone who has undergone any facial surgeries or invasive skin treatments in the last 6 months
* Anyone who is planning to undergo any facial treatments during the study period, including botox, dermal filler, or chemical peels
* Anyone who has not stopped using hormonal birth control within the past month
* Anyone with any chronic skin conditions on the face (e.g., eczema or psoriasis)
* Anyone with a history of skin cancer or pre-cancerous skin lesions on the face
* Anyone currently testing, or plans to in the next 6 weeks, a product for another research study
* Anyone with a history of substance abuse
* Anyone who is currently, or has been for the past 3 months, a smoker
* Anyone with any known allergies or hypersensitivities to any of the study product ingredients:

Truology A2 - Water, Glycerin, Pentylene Glycol, Niacinamide, Cyclodextrin, Polysorbate 20, Squalane, Coco-Caprylate/-Caprate, Cetearyl Alcohol, Cetyl Alcohol, Sodium Hyaluronate, Palmitoyl Tripeptide-5, Caprooyl Tetrapeptide-3, Hydroxyethylcellulose, Ceteareth-20, Beta Glucan, Resveratrol, Dimethyl Sulfone, Retinal, Tocopherol, Tetrahexyldecyl Ascorbate, Dextran, Dipalmitoyl Hydroxyproline, Lactic Acid, Arnica Montana Flower Extract, Glycyrrhiza Glabra (Licorice) Root Extract, Camellia Sinensis (Green Tea) Leaf Extract, Salix Nigra (Willow) Bark Extract, Epilobium Angustifolium Flower/Leaf/Stem Extract, Lonicera Japonica (Honeysuckle) Flower Extract, Lonicera Caprifolium (Honeysuckle) Flower Extract, Rubus Chamaemorus Seed Oil, Sclerotium Gum, Phenoxyethanol, Ethylhexylglycerin, Titanium Dioxide.

C-Boost - Water, Tetrahexyldecyl Ascorbate, Squalane, Glycerin, Propanediol, Caprylic/Capric Triglyceride, Cetearyl Alcohol, Sodium Hyaluronate, Trifluoroacetyl Tripeptide-2, Astaxanthin, Bisabolol, Glutathione, Ergothioneine, Cetearyl Olivate, Sorbitan Olivate, Ceteareth- 20, Dextran, Ferulic Acid, Fulvic Acid, Plankton Extract, Chlorella Vulgaris Extract, Zingiber Officinale (Ginger) Root Extract, Camellia Sinensis (Green Tea) Leaf Extract, Vitis Vinifera (Grape) Seed Extract, Curcuma Longa (Turmeric) Root Extract, Glycyrrhiza Glabra (Licorice) Root Extract, Arctostaphylos Uva-Ursi-Leaf (Bearberry) Extract, Tocopherol, Magnesium Ascorbyl Phosphate, Lecithin, Acrylates/C10-30 Alkyl Acrylate Crosspolymer, Carbomer, Phenoxyethanol, Ethylhexylglycerin, Sodium Hydroxide.

Barrier Restore - *Organic Aloe Barbadensis Leaf Juice, Glycerin, Squalane, Caprylic/Capric Triglyceride, Linoleic Acid, Pentylene Glycol, Cetyl Alcohol, Coco-Caprylate/Caprate, C12-15 Alkyl Benzoate, Cetearyl Alcohol, Fructooligosaccharides, Beta Vulgaris (Beet) Root Extract, Sodium Hyaluronate, Palmitoyl Tripeptide-38, Palmitoyl Tripeptide-5, Palmitoyl Dipeptide-5 Diaminobutyroyl Hydroxythreonine, Palmitoyl Hexapeptide-12, Ceramide Ng, Bisabolol, Tocopherol, Tetrahexyldecyl Ascorbate, Dimethicone, Tetradecyl Aminobutyroylvalylaminobutyric Urea Trifluoroacetate, Tribehenin, Peg 10 Rapeseed Sterol, (Oat) Beta Glucan, Ceteareth-20, Hydroxyethylcellulose, Cetearyl Olivate, Sorbitan Olivate, Hydroxypropyl Cyclodextrin, Cassia Angustifolia Seed Polysaccharide, Linolenic Acid, Tremella Fuciformis Sporocarp Extract, Sarcothalia Circumcincta Extract, Opuntia Ficus-Indica (Nopal Cactus) Extract, Saccharomyces Cerevisiae (Yeast) Extract, Cyathea Medullaris Leaf Extract, Opuntia Streptacantha Stem Extract, Symphytum Officinale (Comfrey) Rhizome/Root Extract, Lycium Chinense (Goji Berry) Extract, Hippophae Rhamnoids (Seabuckthorn) Oil, Lactobacillus Ferment, Acrylates/C10-30 Alkyl Acrylate Crosspolymer, Disodium Edta, Carbomer, Phenoxyethanol, Ethylhexylglycerin, Sodium Hydroxide

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Improvement in self-reported skin health symptoms (measured via questionnaires) | Baseline, Day 1, Week 2, Week 4, Week 6

SECONDARY OUTCOMES:
Changes in overall facial skin quality and health (measured via expert skin grading) | Baseline and Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No